CLINICAL TRIAL: NCT01260298
Title: Protocol To Evaluate Patient Measurements After Ultrasonic Treatment.
Status: Completed | Type: Observational
Sponsor: Sound Surgical Technologies, LLC. (Industry)
Responsible Party: Grant Palmer/Clinical Research, Sound Surgical Technologies, LLC
Other Study IDs: SST2010-2
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Females Scheduled to be Treated Using the MC1.
Keywords: MC1 VASER VASERShape

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MC1 Ultrasonic Device
  Interventions: Device: MC1 Ultrasonic Device

INTERVENTIONS:
Device: MC1 Ultrasonic Device — Ultrasonic and zonal massage device.
  Other Names: MC1; VASERShape

SUMMARY:
The objective of this study is to observe body contour changes following treatment using the MC1 device.

DETAILED DESCRIPTION:
The purpose of this research study is to observe body contour changes following treatment using the MC1 device. The MC1 System is FDA cleared for relief of minor muscle aches, pain and muscle spasm, temporary improvement in local blood circulation, and temporary reduction in the appearance of cellulite.

ELIGIBILITY:
Inclusion Criteria:

1. Is female.
2. Is between 20 and 50 years of age, inclusive, on the day of enrolment.
3. Has a BMI between 20 and 30 kg/m2.
4. Is to be treated in the infra-scapular area using the MC1.
5. Has never been treated with the MC1 before.

Exclusion Criteria:

1. Patient is lactating, has a positive pregnancy test within 7 days of planned study procedure (for female patients of child-bearing potential), or intends to become pregnant during the study or is not using effective methods to prevent pregnancy.
2. Currently enrolled in another device or drug study that has not completed the required follow-up period, or has completed all other study-required follow-up less than 30 days before enrolment in this study.
3. Keloid scars, hypertrophic scars or a history of abnormal healing.
4. Thrombophlebitis.
5. Bleeding or bruising disorders (e.g. idiopathic thrombocytopenic purpura, anticoagulated patients).
6. Tissue ischemia in the area to be treated.
7. Hypertension or abnormally high blood pressure.
8. High cholesterol.
9. Active collagen vascular disease (e.g. fibromyalgia, panniculitis, lupus etc.).
10. Diabetes.
11. Epilepsy.
12. Tuberculosis.
13. Auxiliary electric organs (such as pacemakers), metal or myoelectric prosthesis.
14. Endocrine syndromes or thyroid hyperfunction.
15. Any type of hemorrhagic (bleeding) status.
16. Active skin infection, any infection in the treated area within the last 30 days or skin disease in the area to be treated (e.g. eczema, psoriasis, urticaria, dermographism).
17. Hepatic or renal insufficiency.
18. Bone, muscle or joint disease, dysfunction or healing in the area to be treated.
19. Malignancy in the area to be treated.
20. Laminectomy in the area to be treated. 5.2. Withdrawal and Replacement of Subjects

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female between the ages of 20 and 50 years with BMI between 20 and 30 who are scheduled to be treated using the MC1 device.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kaminer, MD, Principal Investigator — SkinCare Physicians
Locations (1):
- Skin Care Physicians, Chestnut Hill, Massachusetts, United States